CLINICAL TRIAL: NCT00871806
Title: Phase 1, Open-Label, Randomized, Single-Dose, 5-Way Crossover Pilot Bioavailability Study Comparing Eletriptan Oral Disintegrating Tablet Formulations A And B Administered With Or Without Water To Relpax® Commercial Tablets Administered With Water
Brief Title: Pharmacokinetics of Two Eletriptan Oral Formulations Given With and Without Water and the Commercial Tablet Formulation Given With Water
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A1601122
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; eletriptan; bioavailability; oral disintegrating tablet
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Eletriptan commercial tablet with water (Active Comparator): Eletriptan commercial tablet given with water
  Interventions: Drug: Commercial tablet with water
- Eletriptan oral disintegrating tablet (ODT) #1 without water (Experimental): Oral disintegrating tablet formulation #1 without water
  Interventions: Drug: ODT #1 without water
- Oral disintegrating tablet formulation (ODT) #2 without water (Experimental): Oral disintegrating tablet formulation #2 without water
  Interventions: Drug: ODT #2 without water
- Oral disintegrating tablet formulation (ODT) #1 with water (Experimental): Oral disintegrating tablet formulation (ODT) #1 with water
  Interventions: Drug: ODT #1 with water
- Oral disintegrating tablet formulation (ODT) #2 with water (Experimental): Oral disintegrating tablet formulation (ODT) #2 with water
  Interventions: Drug: ODT #2 with water

INTERVENTIONS:
Drug: Commercial tablet with water — 40 mg tablet, given once to each subject
  Arms: Eletriptan commercial tablet with water
Drug: ODT #1 without water — 40 mg tablet given once to each subject
  Arms: Eletriptan oral disintegrating tablet (ODT) #1 without water
Drug: ODT #2 without water — 40 mg tablet given once to each subject
  Arms: Oral disintegrating tablet formulation (ODT) #2 without water
Drug: ODT #1 with water — 40 mg tablet given once to each subject
  Arms: Oral disintegrating tablet formulation (ODT) #1 with water
Drug: ODT #2 with water — 40 mg tablet given once to each subject
  Arms: Oral disintegrating tablet formulation (ODT) #2 with water

SUMMARY:
The study will evaluate whether the blood concentrations of eletriptan administered using two test formulations of oral disintegrating tablets are comparable to those observed with the standard commercial tablet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* No CYP3A4 inhibitors

Exclusion Criteria:

* Clinically significant disease in any organ system
* Positive urine drug screen

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Eletriptan area under the concentration time curve (AUC) and peak concentration (Cmax) | 24 hr

SECONDARY OUTCOMES:
Time of peak eletriptan concentrations (Tmax), half life | 24 hr
Tolerability and safety of treatments assessed by adverse events, vital signs, clinical lab tests | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1601122&StudyName=Pharmacokinetics%20of%20two%20eletriptan%20oral%20formulations%20%20given%20with%20and%20without%20water%20and%20the%20commercial%20tablet%20formulation%20given%20with%20wate